CLINICAL TRIAL: NCT02034942
Title: Substudy of Non-Seda Trial (NCT01967680): Non-sedation Versus Sedation With a Daily Wake-up Trial in Critically Ill Patients Receiving Mechanical Ventilation - Effects on Physical Function. An Investigator-initiated, Randomised, Clinical, Parallel-group, Multinational, Superiority Trial
Brief Title: Non-sedation Versus Sedation With a Daily Wake-up Trial in Critically Ill Patients Receiving Mechanical Ventilation - Effects on Physical Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palle Toft (Other)
Collaborators: Sygehus Lillebaelt (Other); University of Southern Denmark (Other); The Danish Council for Strategic Research (Other)
Responsible Party: Sponsor-Investigator, Palle Toft, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: S-20130025a
Record Dates: First submitted 2014-01-09; First posted 2014-01-14 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Critically Ill; Muscular Atrophy
Keywords: non-sedation
MeSH Terms: conditions — Critical Illness; Muscular Atrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-sedation (Experimental): The experimental group will not receive sedatives. Patients are thoroughly and repeatedly informed by the staff of where they are, what have happened, and what type of treatment they are going to receive.
  Participants will be awake and have a natural sleep rhythm. In case these patients develop and outward delirium, it is necessary to have a nurse or other caregiver at the bedside in order to calm the patient. Patients with delirium will be treated with haloperidol.
  Interventions: Other: Non-sedation
- Sedation with daily wake-up (Active Comparator): The control group will be sedated to Ramsay score 3-4. The first 48 hours the patients will be sedated with propofol, after 48 hours midazolam will be used. During daytime, the patient will be awakened as the intravenous infusion of sedatives will be discontinued. The patient will be considered to be awake when he/she can perform at least three of the following four tasks:
  * Open the eyes to verbal commands.
  * Follow the examiner's instructions with the eyes.
  * Squeeze hands on request.
  * Stick out the tongue on request.
  After a successful wake-up, the infusion of sedative will be resumed, starting on half of the pre-wake-up dose and adjusted to Ramsey score 3-4.
  Interventions: Other: Sedation, control

INTERVENTIONS:
Other: Non-sedation
  Arms: Non-sedation
Other: Sedation, control
  Other Names: Standard treatment, continuous iv-sedation
  Arms: Sedation with daily wake-up

SUMMARY:
Critically ill, ventilator-treated patients rapidly loose much of their muscle mass and strength. This can attribute to prolonged admission, prolonged mechanical ventilation, increased mortality and might have a negative impact on the physical function, degree of independence and quality of life. The pathophysiological background for the loss of muscle mass as well as possible effective treatment is still not well established. In the NONSEDA-trial we randomise critically ill patients to non-sedation or sedation with a daily wake-up trial during mechanical ventilation in the intensive care unit (ICU). It has never been assessed whether non-sedation reduces the loss of muscle mass and strength.

Aim: To assess the effects of non-sedation versus sedation with a daily wake-up trial on physical function after discharge from ICU.

Hypothesis: that non-sedation during ventilator-treatment will improve the physical function after ICU-discharge, compared with standard treatment of sedation with a daily wake-up.

ELIGIBILITY:
Inclusion Criteria:

* Endotracheally intubated
* Expected time on ventilator > 24 hours
* Age ≥ 18 years
* Informed consent

Exclusion Criteria:

* Severe head trauma where therapeutic coma is indicated
* Therapeutic hypothermia where therapeutic coma is indicated
* Status epilepticus where therapeutic coma is indicated
* Patient has participated in the study before
* Patient is transferred from another ICU with length of stay > 48 hours
* Patient is comatose at admission
* PaO2/FiO2 ≤ 9, if sedation is necessary for oxygenation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Physical function | 3 months after ICU-discharge
  Co-primary outcome of: patient-reported quality of life, as measured by SF-36v2, physical component and degree of independence in activities of daily living, as measured by Barthel Index.
  Since this is a co-primary outcome, the type I error probability associated with the test of the null hypothesis should be less than 0,025.

SECONDARY OUTCOMES:
6 minute walk | 3 months after ICU-discharge
  Walking distance in the 6 minute walk test at 3 months follow-up
Handgrip | 3 months after ICU-discharge
  Handgrip-strength at 3 month follow-up
Thigh muscle size | 3 months after ICU-discharge
  Muscle size, measured as cross section area of the rectus femoris muscle at 3 months follow-up
Biomechanical data | 3 months after ICU-discharge
  Muscle strength, measured using biomechanical measurements - Maximal voluntary contraction (MVC), rate of force developement (RFD) and endurance at 25% of MVC at 3 months follow-up

OTHER OUTCOMES:
Biomechanical data | Within 24 hours of ICU-discharge
  Muscle strength - Maximal voluntary contraction (MVC), rate of force developement (RFD) and endurance at 25% of MVC at ICU-discharge.
Handgrip | Within 24 hours of ICU-discharge
  Handgrip-strength at ekstubation and at ICU-discharge.
Thigh muscle size | Within 24 hours of ICU-discharge
  Muscle size, measured as cross section area of the rectus femoris muscle at ekstubation and at ICU-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Helene K Nedergaard, MD, Principal Investigator — Lillebaelt Hospital, Kolding
Locations (1):
- Lillebaelt Hospital, Kolding, Kolding, Denmark

REFERENCES:
- [Background] Strom T, Martinussen T, Toft P. A protocol of no sedation for critically ill patients receiving mechanical ventilation: a randomised trial. Lancet. 2010 Feb 6;375(9713):475-80. doi: 10.1016/S0140-6736(09)62072-9. Epub 2010 Jan 29. PMID 20116842
- [Derived] Nedergaard HK, Jensen HI, Olsen HT, Strom T, Lauridsen JT, Sjogaard G, Toft P. Effect of non-sedation on physical function in survivors of critical illness - A substudy of the NONSEDA randomized trial. J Crit Care. 2021 Apr;62:58-64. doi: 10.1016/j.jcrc.2020.11.017. Epub 2020 Nov 24. PMID 33276294
- [Derived] Nedergaard HK, Jensen HI, Lauridsen JT, Sjogaard G, Toft P. Non-sedation versus sedation with a daily wake-up trial in critically ill patients receiving mechanical ventilation--effects on physical function: study protocol for a randomized controlled trial: a substudy of the NONSEDA trial. Trials. 2015 Jul 23;16:310. doi: 10.1186/s13063-015-0856-1. PMID 26201718